CLINICAL TRIAL: NCT03055104
Title: Management and Treatment of Patients With Severe Malnutrition in Intensive Care Unit: a Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qinggang GE, M.D. Chief physician, Peking University Third Hospital
Other Study IDs: SeNutri-01
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Severe Malnutrition
Keywords: severe malnutrition; Critically Ill; refeeding syndrome; guideline
MeSH Terms: conditions — Malnutrition; Critical Illness; Refeeding Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severe malnutrition: Patients with severe malnutrition (BMI<13 kg/m2), admitted to Peking University Third Hospital from JAN 2008 are involved in this study. After admission, a multidisciplinary team, consisting of specialists in the field of intensive care, pharmacy, psychology, and physical therapy assessed all patients. Management and treatment of these patients are in accordance with guideline for the management of severe malnutrition in PUTH.
  Interventions: Other: management of severe malnutrition

INTERVENTIONS:
Other: management of severe malnutrition — multidisciplinary assessment; guideline for the management of severe malnutrition in PUTH

SUMMARY:
Severe malnutrition can be seen as a low BMI, great weight loss, and even low levels of micronutrients. Current studies on severe malnutrition are mainly in patient with anorexia nervosa. The refeeding phase of these high-risk patients bears a further threat to health and potentially fatal complications (such as refeeding syndrome, infection and severe arrhythmia). The objective of this study is to investigate complications due to refeeding of patients with severe malnutrition, as well as their mortality rate, establish and modify the guideline for management of severe malnutrition in Peking University Third Hospital.

DETAILED DESCRIPTION:
Severe malnutrition can be seen as a low BMI, great weight loss, and even low levels of micronutrients. Current studies on severe malnutrition are mainly in patient with anorexia nervosa. The refeeding phase of these high-risk patients bears a further threat to health and potentially fatal complications (such as refeeding syndrome, infection and severe arrhythmia).

Intensive care unit of Peking University Third Hospital (PUTH) has treated several patients with severe malnutrition successfully since 2008. Most of these patients had a BMI < 10 (kg/m2) at admission. After admission, a multidisciplinary team, consisting of specialists in the field of intensive care, pharmacy, psychology, and physical therapy assessed all patients. Most of the treatment has been regarded successful with a significant BMI gain and little in-hospital mortality. Based on long-term clinical experience, as well as on evidence-based literature, PUTH nutrition group developed a guideline version 1.0 for the treatment of severe malnutrition in August, 2015.

The objective of this study is to investigate complications due to refeeding of patients with severe malnutrition, as well as their mortality rate, establish and modify the guideline for management of severe malnutrition in PUTH.

This is a single-center, ambispective cohort study. Patients who meet the inclusion and exclusion criteria will be included in our registry. As a non-intervention study, these information as below will be collected: reason for admission, relevant medical history, basic demographic characteristics,anthropometric and clinical data, specific nutrition support regimen and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe malnutrition, admitted to PUTH from JAN 2008. (Severe malnutrition is defined as a body mass index (ratio of weight in kg divided by height in m2) < 13)
* Management and treatment are in accordance with guideline version 1.0 for the treatment of severe malnutrition in PUTH.
* Patients requiring intensive care unit management who developed life-threatening complications (such as severe fluid/electrolyte disorders, severe arrhythmia) or had single-organ/multiorgan dysfunction.

Exclusion Criteria:

* Presence of malignancy.
* Life expectancy of less than 24 hours
* Presence of advanced Acquired Immunodeficiency Syndrome (AIDS)
* Aged < 16 years

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients with severe malnutrition (BMI < 13 kg/m2), admitted to PUTH from JAN 2008 are involved in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
28-day change of BMI | from admission to 28-day/discharge, an average of length of ICU stay is 28-day
All-cause 28-day mortality | from admission to 28-day

SECONDARY OUTCOMES:
The rate of infection in ICU | from admission to discharge of ICU, an average of length of ICU stay is 28-day
The rate of refeeding syndrome | from admission to discharge, an average of length of ICU stay is 28-day
The rate of complications | from admission to discharge, an average of length of ICU stay is 28-day
Length of ICU stay | from admission to discharge of ICU, an average of length of ICU stay is 28-day
Cost-effectiveness of treatment | from admission to discharge of ICU (an average of length of ICU stay is 28-day), from admission to discharge of hospital (an average of length of hospital stay is three-month)
  The outcome is the incremental cost of preventing one treatment failure of refeeding syndrome, infection, and all-cause mortality.
All-cause mortality within six month | from admission to six month
Length of hospital stay | from admission to discharge of hospital, an average of length of hospital stay is three-month

CONTACTS AND LOCATIONS:
Overall Officials: Qinggang Ge, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown C, Mehler PS. Medical complications of anorexia nervosa and their treatments: an update on some critical aspects. Eat Weight Disord. 2015 Dec;20(4):419-25. doi: 10.1007/s40519-015-0202-3. Epub 2015 Jul 3. PMID 26138740
- [Result] Wassif WS, McLoughlin DM, Vincent RP, Conroy S, Russell GF, Taylor NF. Steroid metabolism and excretion in severe anorexia nervosa: effects of refeeding. Am J Clin Nutr. 2011 May;93(5):911-7. doi: 10.3945/ajcn.111.012666. Epub 2011 Mar 2. PMID 21367953
- [Result] Aguera Z, Romero X, Arcelus J, Sanchez I, Riesco N, Jimenez-Murcia S, Gonzalez-Gomez J, Granero R, Custal N, Montserrat-Gil de Bernabe M, Tarrega S, Banos RM, Botella C, de la Torre R, Fernandez-Garcia JC, Fernandez-Real JM, Fruhbeck G, Gomez-Ambrosi J, Tinahones FJ, Crujeiras AB, Casanueva FF, Menchon JM, Fernandez-Aranda F. Changes in Body Composition in Anorexia Nervosa: Predictors of Recovery and Treatment Outcome. PLoS One. 2015 Nov 23;10(11):e0143012. doi: 10.1371/journal.pone.0143012. eCollection 2015. PMID 26600309
- [Result] Practice guideline for the treatment of patients with eating disorders (revision). American Psychiatric Association Work Group on Eating Disorders. Am J Psychiatry. 2000 Jan;157(1 Suppl):1-39. No abstract available. PMID 10642782
- [Result] National Collaborating Centre for Mental Health (UK). Eating Disorders: Core Interventions in the Treatment and Management of Anorexia Nervosa, Bulimia Nervosa and Related Eating Disorders. Leicester (UK): British Psychological Society (UK); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK49304/ PMID 23346610
- [Result] Hebebrand J, Himmelmann GW, Herzog W, Herpertz-Dahlmann BM, Steinhausen HC, Amstein M, Seidel R, Deter HC, Remschmidt H, Schafer H. Prediction of low body weight at long-term follow-up in acute anorexia nervosa by low body weight at referral. Am J Psychiatry. 1997 Apr;154(4):566-9. doi: 10.1176/ajp.154.4.566. PMID 9090350
- [Result] Vignaud M, Constantin JM, Ruivard M, Villemeyre-Plane M, Futier E, Bazin JE, Annane D; AZUREA group (AnorexieRea Study Group). Refeeding syndrome influences outcome of anorexia nervosa patients in intensive care unit: an observational study. Crit Care. 2010;14(5):R172. doi: 10.1186/cc9274. Epub 2010 Sep 28. PMID 20920160
- [Result] Hofer M, Pozzi A, Joray M, Ott R, Hahni F, Leuenberger M, von Kanel R, Stanga Z. Safe refeeding management of anorexia nervosa inpatients: an evidence-based protocol. Nutrition. 2014 May;30(5):524-30. doi: 10.1016/j.nut.2013.09.019. Epub 2014 Jan 29. PMID 24698345
- [Result] Saito S, Kobayashi T, Kato S. Management and treatment of eating disorders with severe medical complications on a psychiatric ward: a study of 9 inpatients in Japan. Gen Hosp Psychiatry. 2014 May-Jun;36(3):291-5. doi: 10.1016/j.genhosppsych.2014.02.001. Epub 2014 Feb 10. PMID 24630897